CLINICAL TRIAL: NCT03218384
Title: Ferric Carboxymaltose to Improve Skeletal Muscle Metabolism in Heart Failure Patients With Functional Iron Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to complete enrollment as planned.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-00444
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Results first posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Iron-deficiency
Keywords: Injectafer; ferric carboxymaltose; Supplemental Iron
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ferric Carboxymaltose (Experimental): HF patients with functional iron deficiency assigned to receive one-time dose of Ferric Carboxymaltose 750 mg. Participants will undergo serial assessment before and 4 weeks after study drug administration
  Interventions: Drug: Ferric Carboxymaltose; Device: 31P MRS/MRI
- Placebo (Active Comparator): HF patients with functional iron deficiency assigned to receive one-time dose of Placebo (saline injection). Participants will undergo serial assessment before and 4 weeks after study drug administration.
  Interventions: Drug: Placebo; Device: 31P MRS/MRI

INTERVENTIONS:
Drug: Ferric Carboxymaltose — Intravenous Ferric Carboxymaltose 750 mg mixed under sterile conditions in 100 ml of normal saline for final concentration of 7.5 mg/ml and administered via volumetric infusion pump over 15 minutes.
  Other Names: Injectafer
  Arms: Ferric Carboxymaltose
Drug: Placebo — 100 ml of normal saline solution, and administered via volumetric infusion pump over 15 minutes.
  Other Names: Saline
  Arms: Placebo
Device: 31P MRS/MRI — Each participant will perform the same rhythmic plantar extension exercise protocol twice, for sequential acquisition of magnetic resonance spectroscopy (MRS) and magnetic resonance imaging (MRI) measurements. For the exercise protocol, the participant will lay supine on the scanning table with the right leg inside the volume coil. The exercise consists of repeated plantar flexion movements using resistance bands at a frequency of one repetition per second for 1-2 minutes. Data are collected continuously for 2 minutes before the exercise (baseline), during exercise, and 5 minutes after the exercise for the MRS and MRI experiments.
  Other Names: 3T Siemens MRI

SUMMARY:
The purpose of this study is to better understand how body levels of iron affect the ability to exercise in patients with heart failure (HF).

Heart failure is a condition in which abnormal pumping action of the heart reduces the flow of blood to the body. Patients with heart failure may feel shortness of breath or leg fatigue when they exercise. Iron is an essential nutrient in the diet. In heart failure patients, low body levels of iron might increase shortness of breath and fatigue.

DETAILED DESCRIPTION:
The purpose of this prospective, double blind parallel group randomized study is to compare the effects of ferric carboxymaltose vs. placebo on skeletal muscle mitochondrial oxidative capacity, submaximal exercise tolerance, and health-related quality of life in non-anemic Heart Failure (HF) patients with functional iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic NYHA Class II-III heart failure >3 months
* Guideline-recommended heart failure treatment for > 3 months
* Hemoglobin >13 g/dl for men and >12 g/dl for women
* Functional iron deficiency (defined as serum ferritin level <100 ng/ml or between 100 and 299 ng/ml with transferrin saturation <20%)
* Left ventricular ejection fraction <40%, or left ventricular ejection fraction ≥40% with left atrial enlargement (left atrial volume index >28 ml/m2) and/or left ventricular hypertrophy (left ventricular mass index >95 g/m2 (women) or >115 g/m2 (men) determined by echocardiogram within last 24 months.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Presence of implantable defibrillator, permanent pacemaker, other metal implant not compatible with 3TMRS/MRI, or other contraindication to 3T MRS/MRI procedures
* Heart failure due to infiltrative cardiomyopathy, restrictive cardiomyopathy, or hypertrophic cardiomyopathy
* Weight <50 kg or >120 kg
* Coronary or cerebral atherothrombotic events in the past 6 months
* Hospitalization of emergency room visit for heart failure within past 3 months
* ICD shock in last 3 months
* Known peripheral artery disease or ankle-brachial index <0.9 at screening visit
* Exercise primarily limited by angina, lung disease or neuromuscular disease
* Systolic blood pressure <100 or >160 mmHg
* Heart rate <50 or >110 min-1
* Estimated glomerular filtration rate <30 ml/min
* Liver function tests >3 times upper limit of normal
* Serum phosphate below normal limit
* Pregnant or breast-feeding women
* Women of child-bearing potential unwilling to use recommended contraception methods during the study
* Treatment with oral iron supplements (except multivitamins) in past year
* Treatment with intravenous iron in past year
* Treatment with erythropoiesis stimulating agents in the past year
* Known intolerance of intravenous iron
* History of anaphylaxis
* Participation in another clinical trial within last 30 days.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferric Carboxymaltose | Placebo
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.85) | 56.3 (13.61) | 60.67 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-Exercise Phosphocreatine Recovery Time
Description: Post-exercise phosphocreatine recovery time (in seconds) will be used to assess mitochondrial oxidative capacity. It is measured non-invasively with 31P-magnetic resonance spectroscopy.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 2 | 3
seconds | -0.21 (4.66) | -27.26 (49.27)

2. Secondary Outcome: Change From Baseline in 6-Minute Walk Test Distance
Description: The 6-minute walk test measures the distance that a patient can walk on a flat, hard surface in a period of 6 minutes.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 3 | 3
meters | -12.5 (17.4) | 54.6 (29)

3. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire Score
Description: 23-item self-assessment of symptoms, physical and social limitations, and quality of life in patients with heart failure. KCCQ responses are provided along a rating scale continuum with equal spacing from worst to best. The total score ranges from 0-100, with higher scores indicating better health status. An increase in scores indicates health status improved during the observational period.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 8.7 (13.3) | 14 (10.6)

4. Secondary Outcome: Change From Baseline in Hemoglobin Levels
Description: Hemoglobin is a protein in red blood cells that carries oxygen. Hemoglobin levels (g/dL) were measured in laboratory analyses using patient blood samples.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: Hemoglobin levels (g/dL)
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 3 | 3
Hemoglobin levels (g/dL) | -0.2 (0.4) | 0.1 (0.6)

5. Secondary Outcome: Change From Baseline in Serum Ferritin Levels
Description: Ferritin is a blood protein that contains iron. Serum ferritin levels (ng/ml) were measured in laboratory analyses using patient blood samples.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: Serum ferritin levels (ng/ml)
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 3 | 3
Serum ferritin levels (ng/ml) | 299.7 (118.1) | 2 (7.2)

6. Secondary Outcome: Change From Baseline in Transferrin Saturation
Description: Transferrin saturation, measured as a percentage, is the value of serum iron divided by the total iron-binding capacity of the available transferrin. Transferrin saturation was measured in laboratory analyses using patient blood samples.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 3 | 3
percent (%) | 10.5 (10) | 0.3 (5.1)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Non-systematic assessment- self-reporting by participant
Arm/Group | Ferric Carboxymaltose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (N=3) | Placebo (N=3)
Right buttock pain radiating through leg (Injury, poisoning and procedural complications) | 0 | 1
Hip pain (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03218384/Prot_SAP_000.pdf